CLINICAL TRIAL: NCT01145183
Title: H-26605: Pharmacogenetics of Doxazosin for Cocaine Dependence
Brief Title: Pharmacogenetics of Doxazosin for Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Waggoner Chair and Professor of Psychiatry, Neuroscience, Pharmacology, Immunology and Pathology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: P50DA018197-05 (NIH); P50DA018197-05 (NIH); P50DA018197 (NIH); DPMC (Registry Identifier: NIDA)
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Dependence; Substance Related Disorders; genotype
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxazosin (Experimental): Doxazosin is a long-acting and selective alpha 1-NE blocker, which inhibits the binding of norepinephrine to alpha receptors in the autonomic nervous system.
  Interventions: Drug: Doxazosin
- Placebo (Placebo Comparator): Matched placebo daily dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxazosin — Doxazosin is initiated at 4 mg/wk, and titrated up to a maximum of 8 mg/day over approximately 2 weeks. Participants will be maintained on 6mg-8mg daily dosing until week 13. The subjects will undergo the discontinuation from the study medication during weeks 14 -15.
  Other Names: Cardura (Doxazosin Mesylate)
  Arms: Doxazosin
Drug: Placebo — Matched placebo daily dosing
  Other Names: sugarpills ( Capsules)
  Arms: Placebo

SUMMARY:
Doxazosin, an alpha 1-adrenergic receptor antagonist, may play an important role in cocaine addiction in humans. This study will evaluate to what extent the prospective screening for catecholamine related polymorphisms for alpha 1 NE receptor/transporter, COMT and DBH as main targets predict the treatment efficacy of doxazosin for cocaine-using behavior.

DETAILED DESCRIPTION:
The NE system, especially the alpha 1-adrenergic receptor, may play an important role in cocaine addiction in humans. The results of this study will provide medical safety data on the duration of the induction schedule that will be optimal for attaining our target dose of 8 mg doxazosin daily and will guide future pharmacotherapy trials using Doxazosin or related alpha 1 receptor antagonists for cocaine addiction.

This 16-week double-blind, placebo controlled clinical trial will provide treatment for 100 cocaine-dependent patients and includes a 13 week medication trial (weeks 1-13) and up to 2 week washout period(weeks 14-15). Qualifying subjects will be randomized to receive Doxazosin 8 mg/day, or placebo during the study participation.

Subjects will be receiving 1 mg study medication/placebo capsules at week 1, with 4mg/week induction rate for weeks, according to their randomized assignments, and are maintained on these agents through week 13. At the end of the study (weeks 14-15), participants will undergo discontinuation from active/placebo medication over a 2-week period. Subjects who wish to be transferred to an appropriate treatment program or treatment-research program will be helped with referral during the 2 week period (weeks 14-15).

ELIGIBILITY:
Inclusion Criteria: (1) Signed informed consent form (2) Subject understands the risk and benefits and agrees to visit frequency and procedures (3) Male or female (4) Any race or ethnic origin (5)Diagnosis of cocaine-dependence according to DSM-IV criteria (6) between the ages of 18 and 64 (7)Must be current users of cocaine with self-reported use of cocaine at least once weekly for at least one month preceding study entry, cocaine-positive urine screen and score over 3 which is the cut-off for diagnosis of cocaine dependence as assessed with the Severity of Dependence Scale (Kaye & Darke 2002; Gossop, et al 1995; Gossop, et al. 1997) (8)Women of childbearing age are eligible to be included in the study if they have a negative pregnancy test at screening, agree to adequate contraception to prevent pregnancy, to have monthly pregnancy tests, and they understand the risk of fetal toxicity due to medication.

Exclusion Criteria: (1)Current diagnosis of other drug , especially alcohol or benzodiazepine dependence or abuse (other than cocaine or tobacco) (2) Significant medical conditions (e.g., major cardiovascular, renal, endocrine, hepatic disorders) such as abnormal liver function (with laboratory findings of SGOT or SGPT greater than three times normal), hypotension or hypertension, a current cardiac condition, and those having a high risk of cardiovascular disease, seizure disorders, or another significant underlying medical condition which would contraindicate Doxazosin treatment (3)Lifetime schizophrenia, bipolar disorder, or other psychotic disorders (4) Actively considering plans of suicidality or homicidality (5) Current use of a prescribed psychotropic medication that cannot be discontinued (6) Women planning to become pregnant or breastfeed during the study, or refuse to use a reliable form of birth control or refuse monthly pregnancy testing (7) Subjects who are prescribed any anti-hypertension drugs, except thiazides, will be excluded because these medications may interact with Doxazosin's brain effects in reducing cocaine abuse.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 201 individuals seeking treatment for cocaine dependence were screened between October 2009 and September 2013 at the Outpatient Clinical Trials Research Clinic at MEDVAMC. 16 participants were excluded because they did not meet the inclusion criteria, and 89 participants were lost to follow up before randomization into this study.
Pre-assignment Details: Thus, 96 individuals entered into the study and were randomly assigned into the doxazosin or the placebo groups. Following randomization, 7 participants were lost to follow up and 13 opted out of the pharmacogenetic testing. In total, 76 CUD patients participated in this trial.
Groups:
- Doxazosin (AA Genotype); Doxazosin (AT/TT Genotype): A single dose of doxazosin (8 mg/day) was used in the active medication arm with titration up to 8 mg occurring over a 2-week period.
- Placebo (AA Genotype); Placebo (AT/TT Genotype): Matched placebo daily dosing
Period: Overall Study
Arm/Group | Doxazosin (AA Genotype) | Doxazosin (AT/TT Genotype) | Placebo (AA Genotype) | Placebo (AT/TT Genotype)
Started | 21 | 26 | 19 | 10
Completed | 21 | 26 | 19 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxazosin (AA Genotype) | Doxazosin (AT/TT Genotype) | Placebo (AA Genotype) | Placebo (AT/TT Genotype) | Total
Number analyzed (Participants) | 21 | 26 | 19 | 10 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 26 | 19 | 10 | 76
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (6) | 48.9 (10.2) | 46.6 (9.2) | 48.8 (6) | 48 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 5 | 2 | 20
  Male | 15 | 19 | 14 | 8 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 19 | 16 | 5 | 55
  White | 6 | 7 | 3 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 26 | 19 | 10 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cocaine Positive Urine Toxicology
Description: Cocaine positive urines
Time Frame: 2 weeks blocks throughout study
Measure: Number; unit: percentage of positive urines
Arm/Group | Doxazosin (AA Genotype) | Doxazosin (AT/TT Genotype) | Placebo (AA Genotype) | Placebo (AT/TT Genotype)
Number analyzed (Participants) | 21 | 26 | 19 | 10
percentage of positive urines
  Weeks 1-2 | 88.6 | 85.6 | 75.7 | 75.9
  Weeks 3-4 | 88.6 | 84.7 | 82.8 | 84.7
  Weeks 5-6 | 84.9 | 68.0 | 84.9 | 95.7
  Weeks 7-8 | 75.5 | 70.3 | 77.2 | 100.0
  Weeks 9-10 | 86.3 | 61.9 | 80.6 | 97.0
  Weeks 11-12 | 82.8 | 67.3 | 81.2 | 100.0

2. Secondary Outcome: Adverse Events
Description: Adverse effects were closely monitored during each clinic visit throughout this trial. Vital signs including blood pressure (both pre-medication and post-medication) were measured and documented as were concomitant medications.
Time Frame: Pre- and post study medication
Measure: Number; unit: events
Groups:
- Doxazosin: Doxazosin 8 mg/day
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 47 | 29
events | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse effects were closely monitored during each clinic visit throughout this trial. Vital signs including blood pressure (both pre-medication and post-medication) were measured and documented as were concomitant medications.
Arm/Group | Doxazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/29
Other Adverse Events (participants affected / at risk) | 0/47 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes